CLINICAL TRIAL: NCT05467592
Title: Central Sensitization in Patients Seeking Outpatient Physical Therapy Services
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Neena Sharma, PT, PhD, CMPT, Principal Investigator, University of Kansas Medical Center
Other Study IDs: STUDY00148639
Record Dates: First submitted 2022-05-16; First posted 2022-07-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain; Knee Osteoarthritis; Neck Pain
MeSH Terms: conditions — Low Back Pain; Osteoarthritis, Knee; Neck Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard Physical Therapy care — All therapy will be given as it would have routinely been administered in the clinic. Standard care for all patients includes physical therapy and chiropractic treatment at each visit. There is a nurse practitioner on site. If necessary, patients can receive trigger point injections to the musculature around the back and neck, platelet rich plasma, or headache injections by the nurse practitioner. These interventions vary on a case by case basis. Involvement in the study will not impact the patients plan of care. We will collect this information as confounders and factor into statistical analysis.
  Other Names: Physical Therapy

SUMMARY:
This is an observational study to examine presence of CS in patients with knee osteoarthritis (OA), chronic LBP (CLBP), and chronic neck pain (CNP) seeking outpatient physical therapy (PT) services. The study will also examine if outcomes differ between patients with CS and patients without CS symptoms with standard PT interventions.

DETAILED DESCRIPTION:
Central Sensitization (CS), defined as augmented pain processing, is common in subgroup of nearly all chronic pain conditions, including fibromyalgia, CLBP, OA, and chronic tension headache. However, current studies of CS are primarily limited to research settings, lacking the knowledge about prevalence of CS and rehabilitation outcomes in usual clinical care.

Practicing clinicians do not routinely assess for CS symptoms. Without proper screening for CS, and lack of knowledge of varying levels of nervous system involvement contributing to pain, clinicians are unable to fully identify the depth of the mechanisms and therefore unable to fully determine the best treatment strategies. This observational study addresses this gap in knowledge by screening patients for CS symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of knee, neck, or back pain
* Chronic pain as defined pain > 3 months
* Able to read and understand English

Exclusion Criteria:

* Pregnancy
* Pain less than 3 months

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All subjects over the age of 18 with knee OA, CLBP, and CNP will be asked to consent.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with knee OA, CLBP, and CNP presenting with CS symptoms. | Through study completion, up to 16 weeks
  Percentage of patients with knee OA, CLBP, and CNP presenting with CS symptoms.
2011 Fibromyalgia (FM) survey | Through study completion, up to 16 weeks
  A standard questionnaire for centralized pain. Scores 3-6 in widespread pain index and 9 or greater in symptom severity suggest widespread pain
Beck Anxiety Inventory | Through study completion, up to 16 weeks
  A standard questionnaire with 21 questions. Scores 0-21=low anxiety, scores 22-35=moderate anxiety and scores 36 and above=potentially concerning level of anxiety
Pittsburg sleep scale | Through study completion, up to 16 weeks
  A standard questionnaire to examine sleep problems. A total of 5 scores or greater indicate poor sleep quality
Fear Avoidance Questionnaire | Through study completion, up to 16 weeks
  A standard questionnaire to examine fear related to work and physical activities.
Lower Extremity Functional Scale (LEFS) for patients with knee OA | Through study completion, up to 16 weeks
  LEFS is a 20-question survey about the participant's ability to perform everyday tasks.
Neck Disability Index (NDI) for patients with CNP | Through study completion, up to 16 weeks
  NDI is a 10-question survey in which participants check a box corresponding to how their neck pain impacts their activities of daily living.
Oswestry Disability Index (ODI) for patients with CLBP | Through study completion, up to 16 weeks
  ODI is a 10-question survey in which participants check a box corresponding to how their low back pain impacts their activities of daily living.
Physical Therapy examination data | Through study completion, up to 16 weeks
  Routine PT subjective and objective examination data that includes history taking, range of motion, muscle testing, and neurological exam if necessary
Functional Exam as part of routine primary PT | Through study completion, up to 16 weeks
  Routine PT functional assessment includes gait, sit-to-stand, stair climbing, and squats
Neck flexor muscle performance | Through study completion, up to 16 weeks
  Strength and endurance. Strength will be tested manually with 0-5 MMT standard grading scale or with use of dynamometer for strength and endurance performance of individual muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Neena Sharma, Principal Investigator — University of Kansas Medical Center
Locations (1):
- LifeWorks, Shawnee Mission, Kansas, United States

IPD SHARING:
Plan to Share IPD: No